CLINICAL TRIAL: NCT04225520
Title: Assessment of MEchaNical Dyssynchrony as Selection Criterion for Cardiac Resynchronization Therapy
Brief Title: AMEND-CRT: Mechanical Dyssynchrony as Selection Criterion for CRT
Acronym: AMEND-CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Jens-Uwe Voigt, MD, PhD, Principle Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S64188_v4.0
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Left Ventricular Dyssynchrony; Heart Failure; Cardiomyopathy, Dilated; Cardiac Remodeling, Ventricular
Keywords: Cardiac resynchronization therapy; Heart failure; Mechanical dyssynchrony; Echocardiography; Apical rocking; Septal flash; Left ventricle
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Ventricular Remodeling | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment recommendation based on guidelines (Active Comparator): Treatment of the patient assigned to this arm will be based on the current guidelines for CRT implantation, as issued by the European Society of Cardiology. All patients will receive CRT implantation, with bi-ventricular pacing ON.
  Interventions: Device: Cardiac resynchronization therapy ON
- Treatment recommendation based on mechanical dyssynchrony (Experimental): Treatment of the patients assigned to this arm will be based on the presence of mechanical dyssynchrony. All patients will receive CRT implantation. Bi-ventricular pacing will be either turned ON or OFF, based on respectively the presence or absence of mechanical dyssynchrony.
  Interventions: Device: Cardiac resynchronization therapy ON; Device: Cardiac resynchronization therapy OFF

INTERVENTIONS:
Device: Cardiac resynchronization therapy ON — Implantation of a CRT device. Bi-ventricular pacing will be turned ON.
Device: Cardiac resynchronization therapy OFF — Implantation of a CRT device. Bi-ventricular pacing will be turned OFF.
  Arms: Treatment recommendation based on mechanical dyssynchrony

SUMMARY:
Previous experience with cardiac resynchronization therapy (CRT) candidates suggests that selection of these patients can be improved. Current clinical guideline approaches are mainly too unspecific and lead to a high non-responder rate of 30-40%, which causes a burden on health care systems and puts patients at risk of an unnecessary treatment who might benefit more from a conservative approach. Previous work indicated that using the assessment of mechanical dyssynchrony on echocardiography can lower the non-responder rate at least by 50% without compromising sensitivity for detecting amendable patients. The current prospective, randomized, multi-center trial was therefore designed to prove that the characterization of the mechanical properties of the left ventricle can improve patient selection for CRT. Patients will be randomized into one of two study arms: a control study arm with treatment recommendation based on clinical guidelines criteria, or an experimental study arm with treatment recommendation based on the presence of mechanical dyssynchrony. All patients will receive a CRT implantation. In the control study arm, bi-ventricular pacing will be turned on. In the experimental study arm, bi-ventricular pacing will be turned on or off, depending on the presence or absence of mechanical dyssynchrony, respectively. The primary endpoint will be non-inferiority in outcome of a treatment recommendation based on mechanical dyssynchrony, achieved with a lower number of CRT devices implanted, effectively leading to a lower number needed to treat. Outcome measures are the average relative change in continuously measured LVESV per arm and the percentage 'worsened' according to the Packer Clinical Composite Score per arm after 1 year follow-up.

ELIGIBILITY:
(- - - - - - - - - Inclusion Criteria - - - - - - - - -)

The proposed inclusion criteria represent the minimum recommendations for CRT implantation in heart failure patients according to the ESC 2021 guidelines. In addition:

* Patient has a LVEF ≤ 35%
* Patient has a LVEDD ≥ 2.7cm/m² or LVEDD ≥ 50mm (m) and ≥45mm (f)
* Patient has been in a stable medical condition for ≥ 1 month prior inclusion
* Patient underwent complete revascularization in case of ischemia
* Patients is able to understand and willing to provide a written informed consent
* Patient is 18 years or older

(- - - - - - - - - Exclusion Criteria - - - - - - - - -)

Patients with the following conditions will be excluded:

* unreliable left ventricular volume measurements
* severe MR or more than moderate other valvular disease
* pulmonary hypertension, other than secondary to left heart disease
* patient on hemodialysis
* life expectancy < 1 year
* pregnant or breastfeeding

Patients with prior right ventricular pacing between 20% to 80% will be excluded.

Patients with prior right ventricular pacing ≤ 20% or no pacemaker / ICD will be excluded if they have any of the following criteria:

* PR duration > 250ms
* second / third degree atrioventricular block
* intrinsic QRS duration < 130ms
* atrial fibrillation with resting HR < 50/min or > 80/min

Patients with prior right ventricular pacing ≥ 80% will be excluded if they have any of the following criteria:

* sensed AV delay > 250ms
* paced AV delay > 280ms

Patients with a prior pacemaker / ICD scheduled for LBBaP will be excluded regardless of pacing percentage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Volume response and Packer Clinical Composite Score | 12 months follow-up
  Non-inferiority in outcome of a treatment recommendation based on mechanical dyssynchrony, achieved with a lower number of CRT devices implanted, effectively leading to a lower number needed to treat. Outcome measures are the average relative change in left ventricular end-systolic volume and the proportion of patients 'worsened' according to the Packer Clinical Composite Score after 12 months follow-up.

SECONDARY OUTCOMES:
Effect on left ventricular function in both arms | 12 months follow-up
  * ≥ 10% difference in relative change in left ventricular ejection fraction and/or
  * ≥1.5% difference in absolute change in global longitudinal strain and/or
  * improvement in myocardial work from baseline to month 12
Difference in quality of life as measured by the Minnesota Living with Heart Failure questionnaire score and EuroQol 5D index score in both arms | 12 months follow-up
  * ≥ 5 points difference in change on the Minnesota Living with Heart Failure questionnaire score and/or
  * ≥0.08 points difference in change on the EuroQol 5D index score from baseline to month 12
Difference in 6 minute walk test distance in both arms | 12 months follow-up
  ≥ 45 meters difference in change from baseline to month 12
Difference in predictive value for volume response | 12 months follow-up
  ≥15% relative reduction in left ventricular end-systolic volume from baseline to month 12 will be considered as a response
Difference in predictive value for long-term patient outcome in both arms | 1 year, 3 years and 5 years follow-up
  Cox's proportional hazards model:
  * At 1 year for 'worsened' PCCS
  * At 3 and 5 years for cardiovascular mortality and heart failure hospitalization
Difference in long-term patient outcome in both arms | 3 years and 5 years follow-up
  * Kaplan Meier survival analysis for heart failure hospitalization
  * Kaplan Meier survival analysis for cardiovascular mortality
  * Kaplan Meier survival analysis for combined heart failure hospitalization and cardiovascular mortality
  * Kaplan Meier survival analysis for all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Uwe Voigt, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (24):
- Belgium (8):
  - University Hospital Antwerp, Antwerp
  - ZNA Middelheim, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - AZ Maria Middelares, Ghent
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven
  - AZ Damiaan, Ostend
  - AZ Delta, Roeselare
- Dante Pazzanese Institute of Cardiology, São Paulo, Brazil
- France (3):
  - CHRU Brest, Brest
  - Groupements des hôpitaux de l'institut catholique de Lille, Lille
  - CHU Rennes - Pontchaillou Hospital, Rennes
- Germany (3):
  - St. Vinzenz-Hospital, Cologne
  - Universitätsmedizin Rostock, Rostock
  - Universitätsklinikum Würzburg, Würzburg
- Semmelweis University Heart Center, Budapest, Hungary
- Paul Stradins Clinical University hospital, Riga, Latvia
- Poland (3):
  - Poznan University of Medical Sciences, Poznan
  - Klinika Wad Wrodzonych Serca, Warsaw
  - Silesian Center for Heart Diseases, Zabrze
- CHU de São João, Porto, Portugal
- Heart Institute Nicolae Stancioiu, Cluj-Napoca, Romania
- Hospital Clínico de Barcelona, Barcelona, Spain
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Available upon reasonable request after acceptance of publications.